CLINICAL TRIAL: NCT06516887
Title: A Phase Ib/II Open-Label, Dose-Escalation, Safety, Pharmacokinetic, Pharmacodynamic and Efficacy Study of Bemcentinib Plus Pacritinib In Patients With Advanced Lung Adenocarcinoma
Brief Title: Study of Bemcentinib Plus Pacritinib In Patients With Advanced Lung Adenocarcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 24-0020; 5R01CA269766-02 (NIH)
Record Dates: First submitted 2024-07-09; First posted 2024-07-24 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Advanced Lung Adenocarcinoma
MeSH Terms: interventions — bemcentinib; 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Intervention Model Description: Phase 1b of the study will be conducted to establish the maximum tolerable dose, after pharmacokinetic samples from the first 10 subjects have been collected they will commence Cycle 1, Day 1 treatment. Phase 2 will then be enrolled in a single arm comparison study where some patients will be selected to undergo biopsy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pharmacokinetic Phase 1b (PK) Study Cohort (Experimental): Patients will receive bemcentinib and pacritinib in combination from Days 1 to Day 28. PK samples will be collected on Day 1 (pre-dose, 4, 6h), pre-dose Day 2, Day 7 (pre-dose, 4h and 6h post-dose), pre-dose Day 8, pre-dose Day 14, and Day 22 (pre-dose and 6h post-dose) samples. The Day 22 sample will cover the steady state values for both compounds.
  Six dose levels of combination treatments will be considered:
  * Dose level -1: pacritinib 100 mg oral dose (p.o.) daily + bemcentinib 50 mg p.o. daily;
  * Dose level 1: pacritinib 100 mg oral dose (p.o.) twice daily (BID) + bemcentinib 50 mg p.o. daily;
  * Dose level 2: pacritinib 100 mg p.o. BID + bemcentinib 75 mg p.o. daily;
  * Dose level 3: pacritinib 100 mg BID + bemcentinib 100 mg p.o. daily;
  * Dose level 4: pacritinib 200 mg BID + bemcentinib 100 mg p.o. daily;
  * Dose level 5: pacritinib 200 mg BID + bemcentinib 125 mg p.o. daily.
  Interventions: Drug: bemcentinib; Drug: pacritinib
- Phase II Cohort (Experimental): Of these participants taking the Maximum tolerated dose, up to 15 will undergo a biopsy. Progression free survival will be the primary objective of this study phase.
  Interventions: Drug: bemcentinib; Drug: pacritinib

INTERVENTIONS:
Drug: bemcentinib — Bemcentinib has been investigated in a phase I/II clinical trials for solid tumors. Phase I and II clinical studies of BGB324 are ongoing in non-small cell carcinoma, in which combinations with other agents such as Phase I study of docetaxel (NCT02922777), erlotinib (NCT02424617), and pembrolizumab (NCT03184571) are also being investigated. In a phase I dose escalation study of bemcentinib in combination with docetaxel study, patients with treatment naïve, advanced lung adenocarcinoma receive docetaxel 75 mg/m2 given IV every 21 days in combination with bemcentinib. Bemcentinib dose will be escalated in a standard 3+3 fashion until a maximum tolerated dose is determined.
Drug: pacritinib — For use in clinical studies as an oral agent, pacritinib is supplied as size #0 hard gelatin capsules with gray bodies and scarlet caps. Capsules contain 100 mg pacritinib (free base) and the following inactive ingredients: microcrystalline cellulose NF, polyethylene glycol 8000 NF, and magnesium stearate NF. The capsule gelatin is bovine derived. Pharmacies at investigational sites will receive subject-specific bottles containing 120 capsules packaged in 200 mL high-density polyethylene bottles with child-resistant closures.

SUMMARY:
This is a Phase Ib/II, open-label, single institution dose-escalation, safety, pharmacokinetics, pharmacodynamic and efficacy study.

DETAILED DESCRIPTION:
Specific Aim 1. Determine the safety, tolerability and maximum tolerated dose (MTD) of pacritinib in combination with bemcentinib in patients with advanced lung adenocarcinoma. We propose a prospective, open-label, phase Ib trial to evaluate safety, tolerability and MTD of pacritinib (JAK2 inhibitor) in combination with bemcentinib (AXL inhibitor) in patients with treatment refractory lung adenocarcinoma. The primary objectives of the phase Ib study are to determine the maximum tolerated dose (MTD), pharmacokinetics/pharmacodynamics (PK/PD), dose-limiting toxicities (DLTs) and efficacy of oral pacritinib in combination with bemcentinib. This phase Ib part of the study will use a Bayesian Optimal Interval (BOIN)70 design to determine MTD. This Bayesian dose-finding approach combines the ease of implementation of the traditional "3+3" design with the improved performance of more complex model-based designs in terms of accurately identifying the MTD. Compared to the modified probability toxicity interval design, it has a substantially lower risk of overdosing patients and generally has a higher probability of correctly selecting the MTD. In the phase Ib part of the study, subjects with advanced lung adenocarcinoma will be treated with pacritinib in combination with bemcentinib at increasing doses until MTD for combination treatment has been established. Six dose levels of combination treatments will be considered.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically-or cytologically confirmed diagnosis of locally advanced and/or metastatic lung adenocarcinoma (Stage IV/AJCC Edition 8) (any PD-L1 status) without actionable driver mutations, who has failed at least one line of systemic treatment. Patients with locally advanced and/or metastatic lung adenocarcinoma with driver mutation who have failed standard targeted therapies can also be enrolled on this study.
2. Be refractory to, or intolerant of, an established therapy known to provide clinical benefit for their condition. Patients can be eligible for study if they have failed at least one line of treatment.
3. Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as assessed by the investigator. Evaluable disease in phase 1 is allowed.
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 (AppendixH)
5. Life expectancy of at least 3 months
6. Be ≥18 years of age
7. Negative pregnancy test (if female of childbearing potential)
8. Adequate liver function:

   * Total bilirubin <1.5x upper limit of normal (ULN) (<3xULN for subjects with liver metastases)
   * Aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT), alkaline phosphatase <2.5 x ULN.

     * If liver metastases are present, then AST and ALT <5 x ULN is allowed.
9. Adequate renal function with calculated creatinine clearance ≥30 mL/min by Cockcroft-Gault Formula.
10. Adequate hematologic status:

    * Absolute neutrophil count ≥1500 cells/mm3
    * Platelet count ≥100,000 (plt/mm3)
    * Hemoglobin ≥9 g/dL
11. Have no clinically significant abnormalities on urinalysis
12. Have acceptable coagulation status:

    * Prothrombin time (PT) ≤ 1.5 x ULN
    * Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN
13. Be non-fertile or agree to use an adequate method of contraception. Sexually active patients and their partners must use an highly effective method of contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation and for at least 90 days after the last study drug dose. Female patients using hormonal contraceptive agent should use at least one additional non-hormonal method of contraception (e.g., IUD, condom, abstinence). Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
14. Have read and signed the IRB-approved informed consent form prior to any study related procedure. If a patient is re-screened for the clinical trial or a protocol amendment alters the care of an ongoing patient, a new informed consent form must be signed.
15. Patients enrolled in the Expansion Cohort must be willing to consider pre-study and on-study biopsies, if safe and medically feasible, as determined by a board-certified interventional radiologist. Four to eight core samples will be requested at each biopsy timepoint.
16. Patients must be able to swallow and tolerate oral medications.

Exclusion Criteria:

1. History of the following cardiac conditions:

   1. An acute ischemic cardiac event (e.g., myocardial infarction) or hospitalization for unstable angina within 3 months prior to first dose.
   2. Abnormal left ventricular ejection fraction on echocardiography (less than the lower limit of normal for a subject of that age at the treating institution or Grade 2 severity according to the New York Heart Association as defined by symptoms at less than ordinary levels of activity. Echo will only be considered for symptomatic patients with heart disease and concerns for heart failure. The Echo would be ordered by PI as standard of care.
   3. Uncontrolled cardiac disease, including unstable angina, uncontrolled hypertension (i.e., sustained systolic BP >160 mmHg or diastolic BP >90 mmHg), or need to change medication due to lack of disease control within 12 weeks prior to the provision of consent.
   4. History or presence of bradycardia (≤55 bpm) or history of symptomatic bradycardia, left bundle branch block, cardiac pacemaker or significant atrial tachyarrhythmias as defined by the need for treatment.
   5. Presence of any factors that increase the risk for QTc prolongation, e.g., resistant, or inadequately treated heart failure, presence of hypokalemia or hypomagnesemia not corrected by, or not responding to, replacement therapy or inadequately treated hypothyroidism as defined by the thyroid-stimulating hormone not within the expected range of the institution.
   6. Family history of long QTc syndrome or ventricular arrhythmias; personal history of long QTc syndrome or previous drug induced QTc prolongation of at least Grade 3 (QTc >500 ms). (Appendix I)
2. Have a corrected QT interval (QTcF, Fridericia's method) of >450 msec in men and >470 msec in women.
3. Have a seizure disorder requiring anticonvulsants.
4. Presence of symptomatic central nervous system metastatic disease that requires local therapy such as radiotherapy, surgery, or increasing dose of steroids within 2 weeks prior to Day 1 treatment.
5. Have undergone major surgery, other than diagnostic surgery, within 2 weeks prior to Day 1
6. Have active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
7. Are pregnant or nursing.
8. Received treatment with radiation therapy, chemotherapy, or investigational therapy within 28 days or 5 half-lives, whichever occurs first, prior to study entry.
9. Are unwilling or unable to comply with procedures required in this protocol.
10. Have known infection with human immunodeficiency virus, hepatitis B, or hepatitis C. Patients with history of chronic hepatitis that is not active are eligible.
11. Have a serious nonmalignant disease (e.g., hydronephrosis, liver failure (Child Pugh class B or C), or other conditions) that could compromise protocol objectives in the opinion of the clinical investigators.
12. Uncontrolled diarrhea (grade ≥ 2).
13. Recent bleeding (grade ≥2 within the past 3 months unless precipitated by another event (e.g., trauma, surgery).
14. Use of anticoagulant or anti-platelet agents within the prior 14 days other than baby aspirin.
15. Use of strong CYP3A4 inducers or inhibitors within 5 half-lives prior to cycle 1 day 1 treatment. Patients enrolled in PK study should not be taking a moderate/severe CYP3A4 inhibitor or inducer.
16. Are currently receiving any other investigational agent.
17. Have exhibited allergic reactions to a similar structural compound or formulation as pacritinib or bemcentinib.
18. Patients with severe lactose intolerance, hereditary galactose intolerance, LAPP-lactase deficiency and/or glucose-galactose malabsorption at the discretion of the PI>.
19. Have undergone significant surgery to the gastrointestinal tract that could impair absorption or that could result in short bowel syndrome with diarrhea due to malabsorption.
20. Have a history of severe adverse reaction (e.g., hypersensitivity reaction, anaphylaxis) to sulfonamides.
21. Patients who are currently taking H2-receptor agonists (e.g., cimetidine, ranitidine) or proton pump inhibitors (e.g., omeprazole) must be able to discontinue their use at least seven days prior to the first dose of study treatment and throughout the period they are receiving study treatment. Patients who are unable to do so will be deemed ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 48 months
  PFS will be defined as the time from the date of randomization to the date of disease progression or death (any cause), whichever occurs first. Subjects completing study follow-up or initiating a new anticancer therapy prior to documented PD will be censored in the PFS analysis at the last known date the subject was documented progression free prior to completing follow-up or initiating the new therapy.
Overall Response Rate | Up to 48 months
  Overall response rate is defined as the proportion of patients who have a partial or complete response to therapy.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 48 months
  The time from randomization to death from any cause
Clinical Benefit Rate | Up to 48 months
  The percentage of patients with metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No